CLINICAL TRIAL: NCT01951443
Title: Acute Effect of Rg3-enriched Korean Red Ginseng (Steamed Panax Ginseng C.A. Meyer) Standardized Extract on Arterial Stiffness and Aortic and Brachial Blood Pressure in Healthy Individuals
Brief Title: Korean Red Ginseng Rg3 Extract on Arterial Stiffness and Blood Pressure
Acronym: KRAB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: KRAB
Record Dates: First submitted 2013-08-21; First posted 2013-09-26 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-03

CONDITIONS: Arterial Stiffness, Blood Pressure
Keywords: ginseng; clinical trial; vascular; ginsenosides; blood pressure
MeSH Terms: interventions — Asian ginseng; Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ginseng (Experimental): Encapsulated 400mg Rg3-KRG extract
  Interventions: Dietary Supplement: Ginseng
- Wheat Bran (Placebo Comparator): 400mg Wheat Bran capsule
  Interventions: Dietary Supplement: Wheat Bran

INTERVENTIONS:
Dietary Supplement: Ginseng — 400mg of encapsulated Rg3-KRG
  Arms: Ginseng
Dietary Supplement: Wheat Bran — 400mg of encapsulated wheat bran
  Arms: Wheat Bran

SUMMARY:
The purpose of the study is to evaluate the acute effect of a standardized extract of KRG (Rg3-KRG) consisting of 30% total ginsenosides, including 10% Rg3 ginsenoside on arterial stiffness and blood pressure, as measured by the following parameters: aortic augmentation index, peripheral blood pressure, central blood pressure

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age 18-70 years
* BMI < 30 kg/m2
* Brachial systolic blood pressure < 140 mmHg
* Brachial diastolic blood pressure < 90 mmHg

Main Exclusion Criteria:

* BMI >30kg/m2
* Hypertensive (brachial systolic BP ≥140mmHg and/or diastolic BP ≥90mmHg)
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-08; Primary Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the acute effect of Rg3-KRG on arterial stiffness in healthy adult volunteers, as measured by aortic augmentation index (AIx). | Two weeks (measurements taken on two separate visits with minimum one week washout)

SECONDARY OUTCOMES:
To evaluate the acute effect of Rg3-KRG on aortic and brachial blood pressure in healthy adult volunteers. | Two weeks (measurements taken on two separate visits with minimum one week washout)

OTHER OUTCOMES:
To evaluate the acute safety of Rg3-KRG in healthy adult volunteers using a 48hr symptoms questionnaire. | Two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Vladimir Vuksan, PhD, Principal Investigator — Risk Factor Modification Centre - St. Michael's Hospital; Dr. Amir Hanna (Qualified investigator), MD, Principal Investigator — Unity Health Toronto
Locations (1):
- Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada